CLINICAL TRIAL: NCT04243863
Title: A Randomized, Double Blind, Placebo-Controlled, Sequential Group, Dose-Escalation Study to Evaluate the Safety and Pharmacokinetics of Single and Repeat Doses of VNRX-7145 in Healthy Adult Volunteers
Brief Title: VNRX-7145 SAD/MAD Safety and PK in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: VNRX-7145-101; 272201600029C-P00007-9999-2 (NIH); 18-0012 (Other: DMID)
Record Dates: First submitted 2020-01-14; First posted 2020-01-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers
Keywords: VNRX-7145; Safety; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VNRX-7145 (Experimental): Oral dosing
  Interventions: Drug: VNRX-7145
- Placebo (Placebo Comparator): Oral dosing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VNRX-7145 — Part 1: one dose Part 2: 28 doses (once every 8 hour [q8h] dosing for 9 days with a single morning dose on Day 10)
  Arms: VNRX-7145
Drug: Placebo — Part 1: one dose Part 2: 28 doses (once every 8 hour [q8h] dosing for 9 days with a single morning dose on Day 10)
  Arms: Placebo

SUMMARY:
This is a 2-part, first-in-human dose-ranging study to evaluate the safety and pharmacokinetics of escalating doses of VNRX-7145. In part 1, subjects will receive a single dose of VNRX-7145; in part 2 subjects will receive multiple doses of VNRX-7145 for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years
* Males or non-pregnant, non-lactating females
* Body mass index (BMI): ≥18.5 kg/m² and ≤32.0 kg/m²
* Normal blood pressure
* Normal laboratory tests

Exclusion Criteria:

* Current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, autoimmune, hematologic, neoplastic, or neurological disorder
* History of drug allergy
* Abnormal ECG or history of clinically significant abnormal rhythm disorder
* Positive alcohol, drug, or tobacco use/test

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of subjects with adverse events | Day 8
Part 2: Number of subjects with adverse events | Day 17

SECONDARY OUTCOMES:
Part 1: AUC0-tau | Days 1-3
Part 1: Cmax | Days 1-3
Part 1: tmax | Days 1-3
Part 1: CLr | Days 1-3
Part 2: AUC0-tau | Days 1-10
Part 2: Cmax | Days 1-10
Part 2: tmax | Days 1-10
Part 2: CLr | Days 1-10

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Hamed, MD, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (1):
- Worldwide Clinical Trials Early Phase Services, LLC, San Antonio, Texas, United States

REFERENCES:
- [Derived] de Oliveira CF, Dorr MB, van de Wetering J, Lowe K, Sabato P, Winchell G, Chen H, McGovern PC. Safety and pharmacokinetics of single and multiple doses of ledaborbactam etzadroxil with or without ceftibuten in healthy volunteers. Antimicrob Agents Chemother. 2025 Sep 3;69(9):e0021025. doi: 10.1128/aac.00210-25. Epub 2025 Aug 5. PMID 40762486